CLINICAL TRIAL: NCT05425251
Title: Blood Biomarkers to Improve Management of Mild Traumatic BRAIN Injury in the Elderly
Brief Title: BRAINI-2 Elderly Mild TBI European Study
Acronym: BRAINI2ELDER
Status: Completed | Type: Observational
Sponsor: Hospital Universitario 12 de Octubre (Other)
Collaborators: Technical University of Munich (Other); University Hospital, Grenoble (Other); University Hospital, Clermont-Ferrand (Other); Hospital Vall d'Hebron (Other); BioMérieux (Industry); EIT Health (Other)
Responsible Party: Principal Investigator, Alfonso Lagares Gómez-Abascal, Department of Neurosurgery, Head, Hospital Universitario 12 de Octubre
Other Study IDs: HU 12Octubre; EIT-HEALTH 220325 (Other Grant/Funding Number: European Institute of Innovation and Technology - EU co-fund)
Record Dates: First submitted 2022-03-11; First posted 2022-06-21 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Mild Traumatic Brain Injury
MeSH Terms: conditions — Brain Concussion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- BRAINI2-ELDERLY DIAGNOSTIC & PROGNOSTIC: 2370 patients suffering mild Traumatic brain injury
  Interventions: Diagnostic Test: GFAP and UCH-L1
- BRAINI2-ELDERLY REFERENCE: 480 non-tbi elderly reference patients
  Interventions: Diagnostic Test: GFAP and UCH-L1

INTERVENTIONS:
Diagnostic Test: GFAP and UCH-L1 — 2x5mL blood samples will be used to determine the performance of the automated VIDAS TBI platform in assessing serum concentrations of GFAP and UCH-L1 to rule out the need for a CT-scan after mTBI.

SUMMARY:
Mild traumatic brain injury (mTBI) is one of the most frequent emergencies in the elderly population. Despite most mTBI are managed with cranial computed tomography (CT), only 10% of CTs show lesions, determining CT overuse. The use of serum glial fibrillary acidic protein (GFAP) and Ubiquitin C-terminal Hydrolase-L1 (UCH-L1) have shown potential for ruling out the need for cranial CT. However evidence on biomarker use in mild TBI were not based on studies that included aged participants and patients with comorbidities for which biomarker levels could vary. This is why there is a need for a prospective study that assesses the predictive performance of these two biomarkers in the elderly population, both in elderly patients suffering mild TBI and in a reference population, including patients and participants with and without comorbidities.

ELIGIBILITY:
Inclusion Criteria:

* BRAINI2-ELDERLY DIAGNOSTIC & PROGNOSTIC:

  * Patients ≥65 years of age
  * Mild TBI (GCS 13-15 on admission) with indication of brain CT scan in the 12 hours after injury ;
  * Blood sample obtained ≤12 h after injury and CT scan preferably ≤6h from blood sample.
* BRAINI2-ELDERLY REFERENCE:

  * Non TBI patients ≥65 years of age

Exclusion Criteria:

* BRAINI2-ELDERLY DIAGNOSTIC & PROGNOSTIC:

  * Age below 65 years.
  * GCS 3-12 on admission
  * Time of injury unknown
  * Time to injury exceeding 12 hours
  * Primary admission for non-traumatic neurological disorder (e.g., stroke, spontaneous, intracranial hematoma)
  * Penetrating head trauma
  * Patient with mechanical ventilation from the trauma scene or prehospital management.
  * Venipuncture not feasible
  * No realization of brain CT-scan
  * Subject under judiciary control
  * Subject in inclusion period of a drug interventional study
* BRAINI2-ELDERLY REFERENCE:

  * Subject in inclusion period of another drug interventional study
  * Patients harboring a brain tumor
  * Patients that have had a stroke or neurosurgical operation 1 month prior to the inclusion in the study.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: 2370 participants suffering mild TBI; 480 non TBI participants.
Sampling Method: Non-Probability Sample
Enrollment: 2297 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-03-30 (Actual)

PRIMARY OUTCOMES:
Biomarkers diagnostic performance | 12 hours after mild TBI
  Sensitivity, specificity, positive predictive value (PPV) and negative predictive value (NPV) of GFAP and UCHL-1 used separately and in combination to detect the presence or absence of intracranial lesions on CT scan

SECONDARY OUTCOMES:
Determination of the potential of the two biomarkers in predicting neurological symptoms after TBI | 1 week and 3 months
  Early and midterm biomarker predictive performance in terms of predicting neurological outcome. Neurological status at 1 week and 3 months after TBI and Rivermead post concussion questionnaire.
GFAP reference values | 1 Day, day of extraction of the sample
  GFAP serum level distribution in the non-TBI reference population, considering age and comorbidities.
UCHL-1 reference values | 1 Day, day of extraction of the sample
  UCHL-1 serum level distribution in the non-TBI reference population, considering age and comorbidities.
Determination of the potential of the two biomarkers in predicting neurological outcome assessed by the Extended Glasgow Outcome Score (GOSE) after TBI | 1 week and 3 months
  Early and midterm biomarker predictive performance in terms of predicting neurological outcome. Extended Glasgow Outcome Score (GOSE)
Determination of the potential of the two biomarkers in predicting quality of life assessed by Qolibri-OS after TBI | 1 week and 3 months
  Early and midterm biomarker predictive performance in terms of predicting quality of life after mild TBI assessed by Qolibri-OS
Determination of the potential of the two biomarkers in predicting quality of life assessed by EQ-5D-5L after TBI | 3 months
  Midterm biomarker predictive performance in terms of predicting quality of life after mild TBI assessed by EQ-5D-5L
Determination of the potential of the two biomarkers in depression symptoms assessed by PHQ-9 after TBI | 3 months
  Midterm biomarker predictive performance in terms of predicting depression symptoms after mild TBI assessed by PHQ-9

CONTACTS AND LOCATIONS:
Overall Officials: Alfonso Lagares Gómez-Abascal, MD, PhD, Principal Investigator — Hospital Universitario 12 de Octubre
Locations (7):
- France (4):
  - CHU Clermont-Ferrand, Clermont-Ferrand
  - CHU Grenoble-Alpes, Grenoble
  - Hôpital Edouard HERRIOT, Lyon
  - Hôpital Lyon Sud HCL, Lyon
- Klinikum rechts der Isar, Munich, Germany
- Spain (2):
  - Hospital Universitario 12 de Octubre, Madrid, Madrid
  - Hospital Universitari Vall d'Hebron, Barcelona

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lagares A, Payen JF, Biberthaler P, Poca MA, Mejan O, Pavlov V, Viglino D, Sapin V, Lassaletta A, de la Cruz J; Braini2_elderly_investigators Collaborative group. Study protocol for investigating the clinical performance of an automated blood test for glial fibrillary acidic protein and ubiquitin carboxy-terminal hydrolase L1 blood concentrations in elderly patients with mild traumatic BRAIN Injury and reference values (BRAINI-2 Elderly European study): a prospective multicentre observational study. BMJ Open. 2023 Jul 17;13(7):e071467. doi: 10.1136/bmjopen-2022-071467. PMID 37460257